CLINICAL TRIAL: NCT05441943
Title: Lymphaticovenous Anastomosis as a Surgical Treatment for Breast Cancer-Related Lymphedema
Brief Title: Lymphaticovenous Anastomosis as Treatment for Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Caroline Lilja, Principal Investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/59848; S-20210169 (Other: The Research Ethics Committee of the Region of Southern Denmark)
Record Dates: First submitted 2022-06-07; First posted 2022-07-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Lymphedema; Secondary Lymphedema; Iatrogenic Lymphedema; Lymphedema; Lymphedema of Upper Limb; Lymphedema Arm; Lymphedema, Breast Cancer; Breast Neoplasm; Neoplasms; Breast Cancer; Breast Diseases; Lymphatic Diseases; Skin Diseases; Postoperative Complications; Pathologic Processes; Anastomose; Surgery; Surgical; Lymphedema, Postmastectomy; Postmastectomy Lymphedema; Postmastectomy Lymphedema Syndrome Left Upper Limb; Postmastectomy Lymphedema Syndrome Right Upper Limb; Postmastectomy Lymphedema Syndrome
Keywords: Lymphedema; Breast Cancer; Postmastectomy Lymphedema; Lymphoedema; Breast Cancer Lymphedema; Anastomose; Lymphovenous anastomosis; LVA; Surgery; Breast Neoplasm
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms; Neoplasms; Breast Diseases; Lymphatic Diseases; Skin Diseases; Postoperative Complications; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphovenous anastomosis surgery (Experimental): Lymphovenous anastomosis surgery with pre-operative planning using ICG lymphography and ultra high frequency ultrasound.
  Interventions: Procedure: Lymphovenous anastomosis

INTERVENTIONS:
Procedure: Lymphovenous anastomosis — Pre-operative planning prior to lymphovenous anastomosis using ICG lymphography and ultra high frequency ultrasound for mapping of applicable vessels.
  During surgery, mapped vessels are freely dissected and anastomosed.
  Other Names: LVA; Lymphaticovenous anastomosis; Lymphaticovenular anastomosis

SUMMARY:
The primary aim of this study is to investigate and test whether the use of combined indocyanine green (ICG) lymphography and ultra high frequency ultrasonography can correctly identify lymphatic vessels and venoles in close proximity to each other, for identification prior to lymphovenous anastomosis (LVA) surgery.

DETAILED DESCRIPTION:
BACKGROUND

Breast-cancer related lymphedema is a life-disabling side-effect of breast cancer treatment, affecting more than 1 in every 5 patients. With breast-cancer being the most common cancer diagnosis in women, affecting up to 2.3 million new cases globally, and with a generally high survival rate of 80% or higher in developed countries, the number of breast-cancer survivors with long-term sequela is significant. Compression garments have been considered the standard treatment and rehabilitation for lymphedema. Some of the disadvantages with these treatments include variability in patient compliance, clinical effect and lack of statistical significant results. Therefore, the rehabilitation and treatment options for lymphedema are in high demand, affecting patients physical and mental health.

Lymphovenous anastomosis (LVA) surgery is an attempt to re-establish the lymphatic flow, utilizing the patient's own lymphatic- and venous vessels. Surgical treatment seems effective in selective patient groups, but systematic studies for this are lacking. It is based on this lack of knowledge of patient characteristics and preoperative planning that the project's hypothesis and idea was formed.

Indocyanine green (ICG) lymphography is commonly used for identification of lymphatic vessels pre-operatively, and is considered superior to other modalities. However, until recently, the identification of adjacent venoles has remained a challenge. Ultra high frequency ultrasound may have solved the challenge of identifying the small venoles prior to surgery. The combined use of ICG lymphography and ultra high frequency ultrasound may be the key to optimise patient selection and pre-operative planning of lymphovenous anastomosis surgery.

METHOD

This study is designed as a pilot study with a planned inclusion of 10 patients with a 3 months follow-up period.

The inclusion of patients, the surgical procedure and 3 months follow-up evaluation will take place at the Department of Plastic Surgery Odense University Hospital (OUH), Denmark.

The ICG lymphography is performed by injecting ICG subcutaneously, and used for visualization of the superficial lymphatics for preoperative planning. During real-time visualization, lymphatic vessels are drawn up on the patients arm using a permanent marker.

Ultra high frequency ultrasound (>30MHz) has the ability to visualize small, superficial anatomical layers. Using this ultra high frequency ultrasound (70MHz), following the mapped lymphatic vessels, venous vessels are found nearby and likewise mapped for anastomosis.

The number of LVA anastomosis sites is set to a minimum of two sites per extremity. The number of mapped lymphatics vessels and venoles are compared to the number identified during surgery and recorded.

Prior to and 3 months after surgery, patients are seen for objective measures of upper extremity volume, body composition, L-Dex score of the affected arm and health-related quality-of-life, in addition to ICG lymphography.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Iatrogenic lymphedema following treatment for breast cancer in upper extremity
* Possible to obtain informed consent
* Age>18

Exclusion Criteria:

* Duration of disease over 24 months
* Smoker
* Untreated or uncontrolled primary cancer
* No applicable lymphatic vessels identified, using ICG lymphangiography
* No applicable venous vessels identified using ultra high frequency ultrasound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of vessels planned for surgery surgery | Preoperative
  The number of mapped lymphatics vessels and venoles.
Number of vessels found during surgery | Perioprative
  The number of vessels found during surgery. This number will be compared to the number of vessels planned for surgery.

SECONDARY OUTCOMES:
Changes of arm volume | Baseline and 3 months follow-up
  The change of arm volume difference at baseline and at three months follow-up after surgery.
  Volume calculation Manual circumferential measurements are taken from both arms for volume calculation, based on the formula for multiple blunt cones.
  Water displacement for volume assessment The water displacement test estimates the volume of the arm, based on lowering the extremity in a basin of water, and calculating the water volume difference in mL. Both extremities are measured.
Change of extracellular fluid (liters) relative to total body water (liters), measured in percentage. | Baseline and 3 months follow-up
  The change in extracellular fluid (liters), relative to total body water (liters), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Extracellular fluid and total body water measures will be aggregated to one reported value (extracellular fluid (liters) / total body water (liters)).
Changes of intracellular fluid (liters) relative to total body water (liters), measured in percentage. | Baseline and 3 months follow-up
  The change in intracellular fluid (liters), relative to body water (liters), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Intracellular fluid and total body water measures will be aggregated to one reported value (intracellular fluid (liters) / total body water (liters)).
Changes of total body water (liters) relative to weight (kg), measured in percentage. | Baseline and 3 months follow-up
  The change in total body water (liters), relative to body weight (kg), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Total body water and weight measures will be aggregated to one reported value (total body water (liters) / weight (kg)).
Changes of proteins and minerals (kg) relative to weight (kg), measured in percentage. | Baseline and 3 months follow-up
  The change in proteins and minerals (kg), relative to body weight (kg), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Proteins and minerals and weight measures will be aggregated to one reported value (proteins and minerals (kg) / weight (kg)).
Changes of fat mass (kg) relative to weight (kg), measured in percentage. | Baseline and 3 months follow-up
  The change in fat mass (kg), relative to body weight (kg), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Fat mass and weight measures will be aggregated to one reported value (fat mass (kg) / weight (kg)).
Changes in active tissue mass (kg) relative to weight (kg), measured in percentage. | Baseline and 3 months follow-up
  The change in active tissue mass (kg), relative to body weight (kg), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Active tissue mass and weight measures will be aggregated to one reported value (active tissue mass (kg) / weight (kg)).
Changes of skeletal muscle mass (kg) relative to weight (kg), measured in percentage. | Baseline and 3 months follow-up
  The change in skeletal muscle mass (kg), relative to body weight (kg), measured by a stand-on bioimpedance at baseline and 3 months follow-up. The stand-on device measure the body composition through small electric impulses between two electrodes.
  Skeletal muscle mass and weight measures will be aggregated to one reported value (skeletal muscle mass (kg) / weight (kg)).
Changes in L-Dex score | Baseline and 3 months follow-up
  L-Dex score is a measurement of extracellular fluid of the arm. A stand-on bioimpedance device, estimates the extracellular fluid trough electric impulses between its electrodes. Based upon the impedance ratio of the affected and unaffected arm, the bioimpedance calculates a Lymphedema index, called L-Dex ratio score. A number between -10 and 10 is considered normal, and diagnostic for lymphedema if above 10. Its sensitivity and specificity are 0.66 and 0.99, respectively, at a receiver operating characteristic curve (ROC) value of 10. The score correlates with the limb volume and lymphatic function.
Changes in health-related quality-of-life measured by the LYMPH-Q questionnaire | Baseline and 3 months follow-up
  The LYMPH-Q Upper extremity module questionnaire is a validated patient-reported outcome tool for women with breast cancer related lymphedema. The module contains seven individual scales, measuring: symptoms, function, appearance, psychological function, and satisfaction with information on lymphedema and satisfaction with arm sleeve. Each scale gives an independent score reaching from 0 (worst) to 100 (best), which can be used for comparison of change over time. A higher score indicates a better outcome.
  Patients will complete the questionnaire at baseline and 3 months follow-up.
Changes of lymphatic flow pattern before and after surgery by ICG lymphangiography | Baseline and 3 months follow-up
  Video recordings of ICG lymphographies are stored for later classification of the lymphedema. Staging will be done using the MD Anderson scale; a classification system based upon pattern recognition of the dermal backflow from the ICG lymphography, see table 1.
  MD Anderson stage ICG lymphography findings Stage 0 No dermal backflow Stage 1 Many patent lymphatics and minimal dermal backflow Stage 2 Moderate number of patent lymphatics and segmental dermal backflow Stage 3 Few patent lymphatics with extensive dermal backflow Stage 4 Dermal backflow involving the hand Stage 5 ICG does not move proximally to injection site Table 1: MD Anderson classification based upon ICG lymphography findings.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lilja, MD, Principal Investigator — Department of Plastic Surgery at Odense University Hospital; Jens Ahm Sørensen, MD, Prof, PhD, Study Chair — Department of Plastic Surgery at Odense University Hospital; Jørn Bo Thomsen, MD, Prof, PhD, Study Chair — Department of Plastic Surgery at Odense University Hospital
Locations (1):
- Department of Plastic Surgery, Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armer JM, Ballman KV, McCall L, Armer NC, Sun Y, Udmuangpia T, Hunt KK, Mittendorf EA, Byrd DR, Julian TB, Boughey JC. Lymphedema symptoms and limb measurement changes in breast cancer survivors treated with neoadjuvant chemotherapy and axillary dissection: results of American College of Surgeons Oncology Group (ACOSOG) Z1071 (Alliance) substudy. Support Care Cancer. 2019 Feb;27(2):495-503. doi: 10.1007/s00520-018-4334-7. Epub 2018 Jul 6. PMID 29980907
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Maajani K, Jalali A, Alipour S, Khodadost M, Tohidinik HR, Yazdani K. The Global and Regional Survival Rate of Women With Breast Cancer: A Systematic Review and Meta-analysis. Clin Breast Cancer. 2019 Jun;19(3):165-177. doi: 10.1016/j.clbc.2019.01.006. Epub 2019 Jan 29. PMID 30952546
- [Background] Markkula SP, Leung N, Allen VB, Furniss D. Surgical interventions for the prevention or treatment of lymphoedema after breast cancer treatment. Cochrane Database Syst Rev. 2019 Feb 19;2(2):CD011433. doi: 10.1002/14651858.CD011433.pub2. PMID 30779124
- [Background] Drobot A, Bez M, Abu Shakra I, Merei F, Khatib K, Bickel A, Ganam S, Bogouslavski G, Karra N, Mahran B, Kassis W, Kogan L, Drobot D, Weiss M, Koshima I, Kakiashvili E. Microsurgery for management of primary and secondary lymphedema. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):226-233.e1. doi: 10.1016/j.jvsv.2020.04.025. Epub 2020 May 21. PMID 32446874
- [Background] Seki Y, Kajikawa A, Yamamoto T, Takeuchi T, Terashima T, Kurogi N. The dynamic-lymphaticovenular anastomosis method for breast cancer treatment-related lymphedema: Creation of functional lymphaticovenular anastomoses with use of preoperative dynamic ultrasonography. J Plast Reconstr Aesthet Surg. 2019 Jan;72(1):62-70. doi: 10.1016/j.bjps.2018.09.005. Epub 2018 Sep 20. PMID 30292697
- [Background] Brahma B, Putri RI, Reuwpassa JO, Tuti Y, Alifian MF, Sofyan RF, Iskandar I, Yamamoto T. Lymphaticovenular Anastomosis in Breast Cancer Treatment-Related Lymphedema: A Short-Term Clinicopathological Analysis from Indonesia. J Reconstr Microsurg. 2021 Oct;37(8):643-654. doi: 10.1055/s-0041-1723940. Epub 2021 Mar 1. PMID 33648010
- [Background] Wolfs JAGN, de Joode LGEH, van der Hulst RRWJ, Qiu SS. Correlation between patency and clinical improvement after lymphaticovenous anastomosis (LVA) in breast cancer-related lymphedema: 12-month follow-up. Breast Cancer Res Treat. 2020 Jan;179(1):131-138. doi: 10.1007/s10549-019-05450-2. Epub 2019 Sep 21. PMID 31542874
- [Background] Jorgensen MG, Toyserkani NM, Hansen FG, Bygum A, Sorensen JA. The impact of lymphedema on health-related quality of life up to 10 years after breast cancer treatment. NPJ Breast Cancer. 2021 Jun 1;7(1):70. doi: 10.1038/s41523-021-00276-y. PMID 34075045
- [Background] Kibar S, Dalyan Aras M, Unsal Delialioglu S. The risk factors and prevalence of upper extremity impairments and an analysis of effects of lymphoedema and other impairments on the quality of life of breast cancer patients. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12433. Epub 2016 Jan 13. PMID 26764197
- [Background] Ahmed RL, Prizment A, Lazovich D, Schmitz KH, Folsom AR. Lymphedema and quality of life in breast cancer survivors: the Iowa Women's Health Study. J Clin Oncol. 2008 Dec 10;26(35):5689-96. doi: 10.1200/JCO.2008.16.4731. Epub 2008 Nov 10. PMID 19001331
- [Background] Gillespie TC, Sayegh HE, Brunelle CL, Daniell KM, Taghian AG. Breast cancer-related lymphedema: risk factors, precautionary measures, and treatments. Gland Surg. 2018 Aug;7(4):379-403. doi: 10.21037/gs.2017.11.04. PMID 30175055
- [Background] Chang EI, Skoracki RJ, Chang DW. Lymphovenous Anastomosis Bypass Surgery. Semin Plast Surg. 2018 Feb;32(1):22-27. doi: 10.1055/s-0038-1636510. Epub 2018 Apr 9. PMID 29636650
- [Background] Mihara M, Hara H, Araki J, Kikuchi K, Narushima M, Yamamoto T, Iida T, Yoshimatsu H, Murai N, Mitsui K, Okitsu T, Koshima I. Indocyanine green (ICG) lymphography is superior to lymphoscintigraphy for diagnostic imaging of early lymphedema of the upper limbs. PLoS One. 2012;7(6):e38182. doi: 10.1371/journal.pone.0038182. Epub 2012 Jun 4. PMID 22675520
- [Background] Hayashi A, Giacalone G, Yamamoto T, Belva F, Visconti G, Hayashi N, Handa M, Yoshimatsu H, Salgarello M. Ultra High-frequency Ultrasonographic Imaging with 70 MHz Scanner for Visualization of the Lymphatic Vessels. Plast Reconstr Surg Glob Open. 2019 Jan 22;7(1):e2086. doi: 10.1097/GOX.0000000000002086. eCollection 2019 Jan. PMID 30859043
- [Background] Visconti G, Bianchi A, Hayashi A, Salgarello M. Ultra-high frequency ultrasound preoperative planning of the rerouting method for lymphaticovenular anastomosis in incisions devoid of vein. Microsurgery. 2020 Sep;40(6):717-718. doi: 10.1002/micr.30600. Epub 2020 May 5. No abstract available. PMID 32369213
- [Background] Hayashi A, Visconti G, Giacalone G, Hayashi N, Yoshimatsu H. Recent Advances in Ultrasound Technology: Ultra-High Frequency Ultrasound for Reconstructive Supermicrosurgery. J Reconstr Microsurg. 2022 Mar;38(3):193-199. doi: 10.1055/s-0041-1740129. Epub 2021 Dec 17. PMID 34921372
- [Background] Jorgensen MG, Toyserkani NM, Hansen FCG, Thomsen JB, Sorensen JA. Prospective Validation of Indocyanine Green Lymphangiography Staging of Breast Cancer-Related Lymphedema. Cancers (Basel). 2021 Mar 26;13(7):1540. doi: 10.3390/cancers13071540. PMID 33810570
- [Background] Jorgensen MG, Hermann AP, Madsen AR, Christensen S, Sorensen JA. Indocyanine green lymphangiography is superior to clinical staging in breast cancer-related lymphedema. Sci Rep. 2021 Oct 26;11(1):21103. doi: 10.1038/s41598-021-00396-2. PMID 34702877
- [Background] Gupta N, Verhey EM, Torres-Guzman RA, Avila FR, Jorge Forte A, Rebecca AM, Teven CM. Outcomes of Lymphovenous Anastomosis for Upper Extremity Lymphedema: A Systematic Review. Plast Reconstr Surg Glob Open. 2021 Aug 25;9(8):e3770. doi: 10.1097/GOX.0000000000003770. eCollection 2021 Aug. PMID 34476159
- [Background] Visconti G, Hayashi A, Tartaglione G, Yamamoto T, Bianchi A, Salgarello M. Preoperative planning of lymphaticovenular anastomosis in patients with iodine allergy: A multicentric experience. J Plast Reconstr Aesthet Surg. 2020 Apr;73(4):783-808. doi: 10.1016/j.bjps.2019.11.020. Epub 2019 Nov 29. No abstract available. PMID 31813793
- [Background] Gallagher KK, Lopez M, Iles K, Kugar M. Surgical Approach to Lymphedema Reduction. Curr Oncol Rep. 2020 Jul 28;22(10):97. doi: 10.1007/s11912-020-00961-4. PMID 32720071
- [Background] Ogata F, Narushima M, Mihara M, Azuma R, Morimoto Y, Koshima I. Intraoperative lymphography using indocyanine green dye for near-infrared fluorescence labeling in lymphedema. Ann Plast Surg. 2007 Aug;59(2):180-4. doi: 10.1097/01.sap.0000253341.70866.54. PMID 17667413
- [Background] Klassen AF, Tsangaris E, Kaur MN, Poulsen L, Beelen LM, Jacobsen AL, Jorgensen MG, Sorensen JA, Vasilic D, Dayan J, Mehrara B, Pusic AL. Development and Psychometric Validation of a Patient-Reported Outcome Measure for Arm Lymphedema: The LYMPH-Q Upper Extremity Module. Ann Surg Oncol. 2021 Sep;28(9):5166-5182. doi: 10.1245/s10434-021-09887-y. Epub 2021 Jul 5. PMID 34224044
- [Background] Coroneos CJ, Wong FC, DeSnyder SM, Shaitelman SF, Schaverien MV. Correlation of L-Dex Bioimpedance Spectroscopy with Limb Volume and Lymphatic Function in Lymphedema. Lymphat Res Biol. 2019 Jun;17(3):301-307. doi: 10.1089/lrb.2018.0028. Epub 2018 Nov 2. PMID 30388062
- [Background] Mastick J, Smoot BJ, Paul SM, Kober KM, Hamolsky D, Madden LK, Conley YP, Dixit N, Hammer MJ, Fu MR, Miaskowski C. A Comparison of Supine Versus Stand-on Bioimpedance Devices to Assess Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2021 Dec;19(6):553-561. doi: 10.1089/lrb.2020.0058. Epub 2021 Feb 9. PMID 33567232
- [Background] Tang NSJ, Ramakrishnan A, Shayan R. Quality-of-life outcomes after operative management of primary and secondary lymphoedema: a systematic review. ANZ J Surg. 2021 Dec;91(12):2624-2636. doi: 10.1111/ans.16764. Epub 2021 Apr 6. PMID 33825306
- [Background] Karafa M, Karafova A, Szuba A. The effect of different compression pressure in therapy of secondary upper extremity lymphedema in women after breast cancer surgery. Lymphology. 2018;51(1):28-37. PMID 30248729
- [Background] Gasteratos K, Morsi-Yeroyannis A, Vlachopoulos NC, Spyropoulou GA, Del Corral G, Chaiyasate K. Microsurgical techniques in the treatment of breast cancer-related lymphedema: a systematic review of efficacy and patient outcomes. Breast Cancer. 2021 Sep;28(5):1002-1015. doi: 10.1007/s12282-021-01274-5. Epub 2021 Jul 12. PMID 34254232
- [Background] Carl HM, Walia G, Bello R, Clarke-Pearson E, Hassanein AH, Cho B, Pedreira R, Sacks JM. Systematic Review of the Surgical Treatment of Extremity Lymphedema. J Reconstr Microsurg. 2017 Jul;33(6):412-425. doi: 10.1055/s-0037-1599100. Epub 2017 Feb 24. PMID 28235214
- [Result] Fu MR, Cleland CM, Guth AA, Kayal M, Haber J, Cartwright F, Kleinman R, Kang Y, Scagliola J, Axelrod D. L-dex ratio in detecting breast cancer-related lymphedema: reliability, sensitivity, and specificity. Lymphology. 2013 Jun;46(2):85-96. PMID 24354107
- See also: Will, P.A., Wan, Z., Seide, S.E. et al. Supermicrosurgical treatment for lymphedema: a systematic review and network meta-analysis protocol. Syst Rev 11, 18 (2022). https://doi.org/10.1186/s13643-022-01885-9 — https://rdcu.be/cO8Yo

DOCUMENTS (1):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT05441943/Prot_000.pdf